CLINICAL TRIAL: NCT06845215
Title: Comparison of the Efficacy of Transversus Abdominis Plane Block and Erector Spinae Plane Block in Postoperative Analgesia Management After Abdominoplasty
Status: Recruiting | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ERBİL TÜRKSAL, Principal Investigator, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 2012-KAEK-15/2619
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-02

CONDITIONS: Abdominoplasty; Postoperative Pain; Transversus Abdominis Plane (TAP) Block; Erector Spinae Plane Block
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings | interventions — Dental Occlusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients who underwent abdominoplasty and received TAP block: Patients who underwent abdominoplasty and received TAP block for postoperative analgesia, followed by intravenous patient-controlled analgesia (IV PCA).
  Interventions: Procedure: Transversus abdominis plane (TAP) block
- Patients who underwent abdominoplasty and received ESP block: Patients who underwent abdominoplasty and received ESP block for postoperative analgesia, followed by intravenous patient-controlled analgesia (IV PCA).
  Interventions: Procedure: Erector spina plane block (ESP)

INTERVENTIONS:
Procedure: Transversus abdominis plane (TAP) block — Ultrasound-guided TAP block
  Groups: Patients who underwent abdominoplasty and received TAP block
Procedure: Erector spina plane block (ESP) — Ultrasound-guided ESP block
  Groups: Patients who underwent abdominoplasty and received ESP block

SUMMARY:
Introduction: Abdominoplasty involves the removal of excess skin and fat from the abdominal region, rectus sheath plication, and umbilical transposition. The number of cosmetic abdominoplasty procedures has been steadily increasing in recent years. Due to extensive tissue manipulation and large incisions during surgery, postoperative pain has become a significant concern. Studies report that up to 80% of patients experience postoperative pain; however, fewer than half of these patients receive adequate analgesia. Improving postoperative pain control has been shown to facilitate early mobilization, reduce hospital length of stay, lower healthcare costs, and enhance patient satisfaction. Therefore, ensuring effective postoperative analgesia has become a critical aspect of patient management.

Transversus abdominis plane (TAP) block and erector spinae plane (ESP) block are peripheral nerve block techniques that can be used as part of a multimodal analgesia approach for postoperative pain management after abdominoplasty. In this study, we aimed to compare the effects of TAP and ESP blocks on postoperative pain in patients undergoing abdominoplasty.

Aim/Hypothesis:

H0: There is a significant difference in the analgesic efficacy between ultrasound-guided ESP and TAP blocks in postoperative pain management after abdominoplasty.

H1: There is not a significant difference in the analgesic efficacy between ultrasound-guided ESP and TAP blocks in postoperative pain management after abdominoplasty.

Materials and Methods: Our study was designed as a retrospective analysis. Patient records and hospital database will be reviewed to identify all patients who underwent abdominoplasty and received TAP block or ESP block for postoperative analgesia. Demographic data including age, gender, weight, height, body mass index (BMI) and American Society of Anesthesiologists (ASA) classification, as well as comorbidities and medications used will be recorded on case report forms. The type of block performed (TAP or ESP) and postoperative pain scores obtained from pain assessment forms using the Numerical Rating Scale (NRS) at 0, 2, 4, 6, 12 and 24 hours postoperatively will be documented. In addition, data from the patient-controlled analgesia (PCA) device will be recorded, including number of doses demanded (DEM) and number of doses delivered (DEL). Other parameters such as additional analgesic requirements, postoperative nausea and vomiting, itching and patient satisfaction will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent abdominoplasty and received TAP or ESP blocks for postoperative analgesia, followed by monitoring with IV PCA.

Exclusion Criteria:

* Cases in which IV PCA was not used, VAS scoring was unavailable, or complications occurred.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent abdominoplasty in our hospital between July 2018 and July 2023 and met the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | Postoperative 24 hours
  Visual Analogue Scale (VAS). The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Overall Officials: Erbil Türksal, Specialist, Principal Investigator — University of Health Sciences, Ankara Atatürk Sanatorium Training and Research Hospital
Locations (1):
- University of Health Sciences, Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No